CLINICAL TRIAL: NCT05384223
Title: Evaluation of Clinical Effectiveness, Cost, and Implementation Factors to Optimize Scalability of Treatment for Co-occurring SUD and PTSD Among Teens
Brief Title: Evaluation of RRFT for Co-occurring SUD and PTSD Among Teens
Acronym: STAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: University of Colorado, Denver (Other); Indiana University School of Medicine (Other); Oregon Social Learning Center (Other)
Responsible Party: Principal Investigator, Carla Kmett Danielson, Dr. Carla Kmett Danielson, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00113543
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Substance Use Disorders; PTSD
Keywords: Treatment; Adolescent Substance Use; PTSD
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomization will be monitored by the Principal Investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RRFT (Risk Reduction through Family Therapy) (Experimental)
  Interventions: Behavioral: RRFT (Risk Reduction through Family Therapy)
- Treatment as Usual (TAU): Encompass (Active Comparator)
  Interventions: Behavioral: ENCOMPASS (Integrated Treatment for Adolescents and Young Adults)

INTERVENTIONS:
Behavioral: RRFT (Risk Reduction through Family Therapy) — RRFT is an adaptation and integration of existing empirically-supported interventions with similar theoretical rationales targeting similar populations, particularly Multisystemic Therapy principles (MST)for adolescent SUP and Trauma Focused-Cognitive Behavioral Therapy (TF-CBT) components for PTSD in youth. RRFT consists of seven primary components: Psychoeducation and Engagement, Coping, Family Communication, Substance Use, PTSD, Healthy Dating and Sexual Decision-Making, and Revictimization Risk Reduction.
  Arms: RRFT (Risk Reduction through Family Therapy)
Behavioral: ENCOMPASS (Integrated Treatment for Adolescents and Young Adults) — Encompass is currently a research to practice treatment for adolescents with co-occurring substance use disorders and mental health problems and is used as the standard treatment in the target study settings.
  Arms: Treatment as Usual (TAU): Encompass

SUMMARY:
Psychosocial traumatic events during childhood, serve as strong and consistent predictors of substance use problems (SUP) during adolescence and adulthood.PTSD that extends from such trauma often co-occurs with SUP. Despite this well-established link, standard care for adolescents with co-occurring SUP and PTSD for the last several decades has been to treat these problems separately. This compartmentalized approach to treatment creates a burden on teens and families, raises unique challenges to clinicians in both mental health and addiction domains, and may contribute to high rates of SUP relapse among adolescents with co-occurring PTSD. To address this problem, our team recently completed a rigorous National Institute on Drug Abuse (NIDA)-funded randomized controlled trial (RCT) supporting the efficacy of an integrative, exposure-based treatment we developed, Risk Reduction through Family Therapy (RRFT), in greater long term reductions in SUP, as well as PTSD avoidance and hyperarousal symptoms, in comparison to standard treatment in a large teen sample. The proposed RCT, with an effectiveness-implementation Hybrid Type I design, substantially builds on that prior research by proposing to 1) evaluate whether RRFT's clinical effectiveness for reducing SUP and PTSD can be extended to youth in outpatient substance use treatment settings-where youth are presenting for SUP treatment and where clinicians often have less experience treating PTSD (Aim 1); 2)evaluate the cost-effectiveness of RRFT and to explore inner context variables (e.g., perceived treatment acceptability, attitudes, and satisfaction among the participating adolescents, caregivers, agency leaders, and therapists and barriers to and facilitators of implementation) that might affect RRFT implementation in diverse practice settings(Aim 2). The proposed effectiveness-implementation trial will recruit adolescents (13-18 years) with a history of psychosocial trauma presenting with SUP and PTSD symptoms for outpatient substance use disorder treatment at sites in Denver, Colorado. Participants will be randomized to RRFT or Treatment as Usual. A multi-method, multi-respondent approach will track clinical outcomes(SUP, PTSD, and putative targets of treatment, such as emotional suppression)at 3, 6, and 12 months post-baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 13-19 years (adolescents);
2. Experienced lifetime DSM-V PTSD Criteria A-defined potentially traumatic event, such as interpersonal violence, with memory of incident(s), such as child sexual abuse (forced or unwanted vaginal or anal penetration by an object, finger, or penis; oral sex; touching of the respondent's breasts or genitalia; or respondents' touching of another person's genitalia); child physical abuse (nonaccidental physical injury to the child or any action that results in a physical impairment of the child), witnessed domestic violence (exposure to conduct by a household member against another household member that involves attempted or completed assault or murder); witnessed community violence; dating violence; as well as disasters, accidents, etc.;
3. Five or more current DSM-V PTSD symptoms as assessed on the Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS)/UCLA PTSD Index;
4. Substance use, defined as alcohol or non-tobacco drug use, in the past 28 days prior to study screening per self-report. If in a restrictive setting for the 28 days prior to study screening, substance use will be anchored to use prior to entering restrictive setting;
5. A current (past year) non-nicotine substance use disorder (SUD) as assessed on the K-SADS;
6. English-speaking.

Exclusion Criteria:

1. Presence of Pervasive Developmental Disability or Moderate/Severe Mental Retardation or other cognitive limitation that would preclude meaningful engagement in RRFT or cognitive-behavioral therapy
2. Actively suicidal/homicidal;
3. Active psychosis.

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Timeline Follow Back (TFLB) - Change from baseline in # days non-tobacco substance used in past 28 days @ 3,6, and 12 months. | Collected at baseline, 3, 6, & 12 months
  The Timeline Follow Back (TLFB) is a validated, subjective measure that uses a calendar for people to provide estimates of substance use (drugs/alcohol) on a daily basis, retrospectively. Key dates and calendars are used to aid in memory recall. The measure is beneficial in both clinical and research environments. Over time, the TLFB looks for a decrease in substance use. Higher numbers of substance use are indicative of greater substance use.
UCLA PTSD Index DSM V - Change from baseline in UCLA PTSD total score @ 3,6, and 12 months | Collected at baseline, 3, 6, & 12 months
  The University of California, Los Angeles (UCLA) Post Traumatic Stress Disorder Index Diagnostic and Statistical Manuals 4th ed (DSM-IV; UCLA PTSD Index DSM-IV) is a validated, subjective measure that consists of 23 yes or no questions regarding the occurrence of different traumas or losses that may happen during a child's life. Each question is followed up with details of the trauma that occurred and more extensive questioning for the trauma experienced that is still most bothersome in the present day. These follow-up questions gauge symptoms of PTSD on a five-point Likert scale that ranges from "none" (score of 0, no days has this symptom occurred in the last month) to "most" (score of 4, symptom occurred almost every day in the past month). The most traumatic experience is also followed by several yes/no questions that gauge distress and functional impairment. Higher scores are indicative of higher rates of PTSD symptoms.

SECONDARY OUTCOMES:
Urine Drug Screen (UDS) - Between group comparison -total # negative UDS /total # collected at baseline, 3, 6, & 12 months | Collected at baseline, 3, 6, & 12 months
  Participants will complete urine drug screens that will be at least 6 panel including cocaine, THC (tetrahydrocannabinol-marijuana), opiates, amphetamines, methamphetamines, and benzodiazepines
Timeline Follow Back (TFLB) - total # of days/28 day of cannabis use, alcohol use, and other non-nicotine substance use (excluding cannabis, alcohol). | Collected at baseline, 3, 6, & 12 months
  The Timeline Follow Back (TLFB) is a validated, subjective measure that uses a calendar for people to provide estimates of substance use (drugs/alcohol) on a daily basis, retrospectively. Key dates and calendars are used to aid in memory recall. The measure is beneficial in both clinical and research environments. Over time, the TLFB looks for a decrease in substance use. Higher numbers of substance use are indicative of greater substance use.
Response to Stress Questionnaire (RSQ) - Change from baseline in Adolescent/Child's Self-Report Responses to Family Stressors (subscale score items a-l) | Change from baseline @ 3,6, and 12 months
  The RSQ measures coping and involuntary stress responses. Higher scores indicate higher stress.
Alabama Parenting Questionnaire (APQ) - positive parenting subscale, inconsistent discipline subscale, and supervision/monitoring subscale. | Collected at baseline, 3, 6, & 12 months
  The Alabama Parenting Questionnaire (APQ) is a validated measure consisting of questions that look into family interactions and, more specifically, interactions between youth and caregiver. The scale is scored on a five-point Likert scale that ranges from "never" (score of 1) to "always" (score of 5) when looking at how often certain behaviors occur within the home. High scores on the positive parenting subscale and low scores on the poor monitoring/supervision, inconsistent discipline, and corporal punishment subscales are indicative of positive parenting.
Difficulties in Emotion Regulation Scale (DERS) - Change from baseline in total score @ 3, 6, & 12 mo f/u | Change from baseline in total score @ 3, 6, & 12 month follow-up
  The Difficulties in Emotion Regulation Scale (DERS) is an instrument measuring emotion regulation problems. is a 36-item self-report measure of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never") to 5 ("almost always"). Higher scores indicate more difficulty in emotion regulation.
Timeline Follow Back (TLFB) - Average quantity of specific substance used on days of use/28 days | Collected at baseline, 3, 6, & 12 months
  The Timeline Follow Back (TLFB) is a validated, subjective measure that uses a calendar for people to provide estimates of substance use (drugs/alcohol) on a daily basis, retrospectively. Key dates and calendars are used to aid in memory recall. The measure is beneficial in both clinical and research environments. Over time, the TLFB looks for a decrease in substance use. Higher numbers of substance use are indicative of greater substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Kmett Danielson, PhD, Principal Investigator — Medical University of South Carolina; Paula Riggs, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - CU Medicine Psychiatry - Outpatient Clinic, Aurora, Colorado
  - ARTS - Synergy Outpatient Services, Denver, Colorado